CLINICAL TRIAL: NCT05357196
Title: An Open-label Phase I/II Clinical Trial of PT-112 Combine With Gemcitabine Injection for Advanced Solid Tumors
Brief Title: PT-112 (Phosplatin's Platinum) Combine With Gemcitabine Injection for Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-PT112-ONC-P2-002
Record Dates: First submitted 2022-01-13; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Biliary Tract Cancer
Keywords: PT-112
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: One-armed test，An Open-Label Phase I/ II Clinical Study of PT-112 in Combination with Gemcitabine Injection for the Treatment of Patients with Advanced Solid Tumors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PT-112 in Combination with Gemcitabine Injection (Other): PT-112 in combination with Gemcitabine injection for the treatment of patients with advanced solid tumors
  Interventions: Drug: PT-112

INTERVENTIONS:
Drug: PT-112 — Drug: PT-112, The MTD(Maximum Tolerated Dose ) and RP2D of PT-112 when used in combination with gemcitabine will be determined during dose escalation.
  Drug: Gemcitabine, Gemcitabine will be administered at a fixed dose of 1000 mg.
  Other Names: Gemcitabine

SUMMARY:
Phase I dose escalation period: solid tumors, including but not limited to biliary tract cancer, pancreatic cancer, ovarian cancer, thymoma, neuroendocrine carcinoma and other advanced solid tumors.

Phase II trial period: biliary tract cancer

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I/ II clinical study, including phase I dose escalation period and phase II trial period.

The phase I dose escalation period will adopt a 3+3 dose escalation design. Three dose groups are designed as follows:

Level 1: 150 mg/m2 PT-112 (Phosplatin's platinum) + 1000 mg/m2 gemcitabine; Level 2: 200 mg/m2 PT-112 + 1000 mg/m2 gemcitabine; Level 3: 250 mg/m2 PT-112 + 1000 mg/m2 gemcitabine. If any DLT(Dose-Limiting Toxicity ) occurs in Level 1 group during dose escalation, the dose will be down titrated to Level-1 150 mg/m2 PT-112 + 800 mg/m2 gemcitabine. After the lowest dose group (Level-1 or Level 1), the dose of gemcitabine will be fixed while the dose of PT-112 will be up titrated.

During the phase I dose escalation period, sufficient data will be obtained to demonstrate that the dose is safe. Investigators and sponsor will discuss and decide the initiation time of the phase II period. In phase II, it is planned to enroll subjects with biliary tract cancer according to Simon's two-stage study design, to assess the safety and anti-tumor efficacy of PT-112 in combination with gemcitabine for treating patients with advanced biliary tract cancer. In the first period, 23 evaluable subjects are intended to be enrolled. If ≤ 12 subjects have disease control (CR(Complete Response) + PR(Partial Response) + SD(Stable Disease)) at the first post-baseline tumor assessment, the study drug will be considered to be ineffective and the trial terminated; if >12 subjects have disease control (CR + PR + SD), the enrollment for phase II will be initiated. In total, 37 evaluable subjects will be enrolled. The study drug will be considered to be ineffective if a total of ≤23 subjects have disease control (CR + PR + SD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years (18 and 75 years included).
2. For phase I dose escalation period only: patients with locally advanced or metastatic solid tumors (including but not limited to biliary tract cancer, pancreatic cancer, ovarian cancer, etc.) confirmed by histopathology or cytology who have failed to respond to standard regimen or have no standard regimen.
3. ECOG(Eastern Cooperative Oncology Group) performance status score of 0-1.
4. Expected survival time greater than 12 weeks.
5. Subjects must have proper organ function and laboratory test results meet the following standards prior to enrollment:

   * Basically normal bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 × 109/ L, platelet ≥ 100 × 109/ L, and hemoglobin ≥ 90 g/ L;
   * Basically normal liver function: serum albumin ≥ 3.0 g/dL; bilirubin ≤ 1.5 × ULN(upper limit of normal ), ALT(Alanine aminotransferase) and AST( Aspartate transaminase) ≤ 2.5 × ULN; if the patients suffer from liver metastasis or primary liver cancer, ALT or AST ≤ 5 × ULN;
   * Normal renal function: creatinine ≤ 1.5 × ULN or creatinine clearance (CL) ≥ 60 mL/min (according to Cockcroft-Gault formula); .Basically normal coagulation function: INR(international normalized ratio) ≤ 1.5 × ULN, APTT(activated partial thromboplastin time) ≤ 1.5 × ULN.
6. Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%.
7. subjects with a history of brain metastases who are diagnosed as stable disease by the investigator and do not require additional steroids or anticonvulsants, with radiotherapy or without treatment.
8. Negative serum β-HCG(human chorionic gonadotropin) test for women of childbearing potential (defined as women aged less than 50 years or over 50 years and amenorrheic for less than 12 months prior to screening).
9. Subjects must give informed consent for the study prior to the test and sign the informed consent form.

   Additional inclusion criteria applicable to phase II trial period:
10. Patients with histologically or cytologically confirmed unresectable or metastatic biliary tract cancer, including intrahepatic cholangiocarcinoma (IHCC), extrahepatic cholangiocarcinoma (EHCC), and gallbladder carcinoma (GBC).
11. Patients who have not received systemic treatment for unresectable or metastatic biliary tract cancer or received only one systemic anti-tumor chemotherapy regimen; patients who have received one adjuvant or neoadjuvant chemotherapy regimen and relapsed more than 6 months after the end of chemotherapy can be enrolled.

Exclusion Criteria:

1. Positive HIV antibody.
2. Active hepatitis, (hepatitis B: HBsAg positive with abnormal liver function and HBV(hepatitis B virus )-DNA ≥ 1000 IU/ml; hepatitis C: HCV(hepatitis C virus)-RNA positive with abnormal liver function).
3. Treatment with corticosteroids > 20 mg/ day prednisone or other equivalent hormone (unless used to prevent contrast media reactions during radiological procedures), growth factors (eg, erythropoietin, granulocyte colony-stimulating factor, recombinant human thrombopoietin), blood transfusion.
4. The toxic and side effects caused by the subject's previous treatment not recovered to CTCAE Grade ≤ 1, except for alopecia and other events judged to be tolerable by the investigator.
5. Peripheral neuropathy of any grade within 28 days prior to the initiation of study drug.
6. Patients with known sensitivity or hypersensitivity to platinum drugs and/ or gemcitabine.
7. Having received a major surgery within 28 days prior to the initiation of study drug.
8. Having received chemotherapy, biotherapy, radiotherapy, endocrine therapy and targeted anti-tumor therapy (except for nitrosoureas and mitomycin C) within 28 days prior to the initiation of study drug; received nitrosoureas or mitomycin C within 6 weeks prior to the initiation of study drug; received palliative local radiotherapy within 1 week prior to the initiation of study drug; received Chinese herbal medicine with anti-tumor effect within 1 week before the initiation of the study drug.
9. Patients with uncontrollable hypertension (normal range for diastolic blood pressure 60-90 mmHg and for systolic blood pressure 90-140 mmHg ).
10. Requiring systemic treatment for an acute bacterial, viral, or fungal infection, or having an unexplained fever (body temperature > 38.5℃) during screening prior to the first dose.
11. Patients with moderate to large amount of body cavity effusion to be disposed of.
12. With a known history of psychiatric disorders or drug abuse that may affect compliance.
13. Presence of any of the following conditions within 6 months prior to signing informed consent: uncontrolled congestive heart failure (New York Heart Association class II-IV), angina pectoris, myocardial infarction, stroke (except for lacunar infarction), coronary/ peripheral artery bypass graft surgery, pulmonary embolism.
14. Arrhythmia unable to be controlled by drugs or sustained QTc(corrected QT interval ) interval prolongation, > 450 msec in males or > 470 msec in females.
15. Having participated in other clinical studies within 28 days prior to the first dose of the study drug.
16. Pregnant or lactating women.
17. Women of childbearing potential, men of childbearing potential and their partners who are unable to use effective and adequate dual contraception while receiving the study drug and for 3 months after the end of the study.
18. Patient not suitable for participating in the study for any reason judged by the investigator.

    Additional exclusion criteria applicable to phase II trial period:
19. Patients with advanced biliary tract cancer previously treated with gemcitabine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-04-28 (Estimated)

PRIMARY OUTCOMES:
Define the recommended dose level for PT-112(Phase I) | 30 months
  Define the recommended dose level for PT-112, administered on Days 1 and 8 of each 21-day cycle, for pivotal studies based on the risk/benefit ratio of 150 mg/m2 、200 mg/m2 and 250 mg/m2 dose levels.
To obtain best disease control rate (DCR) data(Phase II) | 24 months
  To obtain best disease control rate (DCR) data of 47 subjects who have used PT-112 Injection in combination with Gemcitabine Injection at RP2D(Recommended Phase II Dose ) dose for treating advanced biliary tract cancer. Endpoints: Disease control rate (DCR)

SECONDARY OUTCOMES:
Anti-tumor efficacy evaluation (Phase I) | 30 months
  Disease Control Rate by disease manifestation, evaluated using RECIST 1.1 criteria.
Peak Plasma Concentration (Cmax) (Phase I) | 30 months
  To assess the Peak Plasma Concentration (Cmax) profile of 21 subjects who have used PT-112 in combination with Gemcitabine. PT-112 and Gemcitabine related PK parameters.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability](Phase II) | 24 months
  To obtain the Adverse Events (AEs) of all 47 subjects with advanced biliary tract cancer and have used PT-112 Injection in combination with Gemcitabine Injection for treating . Characterization of the type, incidence, severity, duration, reversibility and relationship to treatment of adverse events (AEs), and effects on vital signs and laboratory parameters.
Area under the plasma concentration versus time curve (AUC) | 30 months
  To assess the Area under the plasma concentration versus time curve (AUC) profile of 21 subjects who have used PT-112 in combination with Gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, M.D., Principal Investigator — Fudan University
Locations (4):
- China (4):
  - ZhongNan Hospital Of Wuhan University, Wuhan, Hubei
  - General Hospital Of Eastern Theater Command, Nanjing, Jiangsu
  - Zhongshan Hospital Fudan Universtity, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital ZheJiang University School Of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No